CLINICAL TRIAL: NCT06414031
Title: Tranexamic Acid for Reduction of Intra- and Postoperative Transfusion Requirements in Elective Abdominal Surgery: Randomized Controlled Trial
Brief Title: Tranexamic Acid for Reduction of Transfusion in Abdominal Surgery
Acronym: TATRA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ulrich Ronellenfitsch, MD (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); Coordinating Centre for Clinical Trials Halle (Unknown)
Responsible Party: Sponsor-Investigator, Ulrich Ronellenfitsch, MD, Professor of Evidence-based Abdominal Surgical Oncology, Martin-Luther-Universität Halle-Wittenberg
Organization: Martin-Luther-Universität Halle-Wittenberg (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TATRA; 01KG2305 (Other Grant/Funding Number: German Federal Ministry of Education and Research); 2023-509970-43-01 (EU CTIS Number)
Record Dates: First submitted 2024-05-10; First posted 2024-05-14 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Surgical Blood Loss; Transfusion-dependent Anemia; Abdomen Disease
MeSH Terms: conditions — Blood Loss, Surgical | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamic acid (Experimental): Intravenous administration of tranexamic acid (1 g bolus 10 minutes prior to skin incision followed by continuous infusion 125 mg / hour until skin closure)
  Interventions: Drug: Tranexamic Acid
- Placebo (Placebo Comparator): Intravenous administration of placebo (normal saline), 50 ml bolus 10 minutes prior to skin incision followed by continuous infusion of 6.25 ml / hour until skin closure.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid — Intravenous administration
  Other Names: Tranexamsäure Carinopharm 100mg/ml
  Arms: Tranexamic acid
Drug: Placebo — Intravenous administration
  Other Names: Isotone Kochsalz-Lösung 0,9% Infusionslösung
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if the administration of tranexamic acid can reduce the necessity of blood transfusions in adult patients undergoing major abdominal surgery. . It will also inform about safety of tranexamic acid in this setting.

The main question it aims to answer is: Does tranexamic acid lower the probability of receiving at least one blood transfusion during or after surgery?

Participants will compare tranexamic acid o a placebo (a look-alike substance that contains no drug) to see if tranexamic acid works to reduce the necessity of a blood transfusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or above
2. Planned elective esophagectomy, gastrectomy, colectomy, rectal resection, pancreatic resection, or hepatectomy
3. Adequate renal function with serum creatinine <250 µmol/L (2.82 mg/dL)
4. Written informed consent obtained before randomization
5. Negative pregnancy test for women of childbearing potential within 14 days of commencing study treatment. Females of reproductive potential must agree to practice highly effective contraceptive measures during the study. These comprise measures with a failure rate of <1% per year when used consistently and correctly, such as intravaginal and transdermal combined (oestrogen and progestogen containing) hormonal contraception, injectable and implantable progestogen-only hormonal contraception, intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion; vasectomised partner, sexual abstinence (defined as refraining from heterosexual intercourse during the entire study period).

Exclusion Criteria:

1. Severe anaemia, defined as a haemoglobin concentration <8 g/dL (<5 mmol/L) or anaemia with haemoglobin concentration ≥8 to <10 g/dL (≥5,0 to <6,2 mmol/l) and one or several of the following symptoms suggesting hypoxemia:

   * Clinical signs of tachycardia, e.g., resting heart rate >100 beats/minute, palpitation etc.
   * Clinical signs of hypotension, e.g., resting systolic blood pressure <100 mmHg, orthostatic dysregulation etc.
   * Clinical signs of dyspnea, e.g., speech dyspnea, resting respiratory rate >20 breaths/min.
2. Thrombocytopenia with platelets <60 x 109 /L
3. Confirmed bleeding disorder with the need for specific preventive perioperative treatment (e.g., factor deficiency with the need of perioperative substitution)
4. A priori refusal of blood transfusions
5. Confirmed thrombophilia with a pertinent need for perioperative anticoagulation
6. Allergy / hypersensitivity to tranexamic acid
7. Recent (<30 days) thromboembolic event
8. History of medically confirmed convulsions
9. In female subjects: pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Transfusion necessity | Until hospital discharge or 30 days postoperatively, whatever occurs earlier
  Intra- or postoperative transfusion of at least one unit of packed red blood cells

SECONDARY OUTCOMES:
Transfusion amount | Until hospital discharge or 30 days postoperatively, whatever occurs earlier
  Number of transfused units of packed red blood cells per patient
Blood loss | From skin incision to suture
  Estimated intraoperative blood loss
Postoperative complications and mortality | Until hospital discharge or 30 days postoperatively, whatever occurs earlier
  Postoperative complications and mortality assessed according to the Clavien-Dindo scheme
Length of hospital stay | From hospital admission to discharge
  Time period from hospital admission to discharge
Operation time | From skin incision to suture
  Time period from skin incision to suture
Anesthesia time | From anesthesia induction to end of anesthesia
  Time period from anesthesia induction to end of anesthesia
D-dimer levels | Until hospital discharge or 30 days postoperatively, whatever occurs earlier
  Serum levels of D-dimers
Adverse events | Until hospital discharge or 30 days postoperatively, whatever occurs earlier
  Any adverse event attributed to the intervention comprising anaphylaxis, thromboembolic events, acute renal failure, acute heart failure, seizures

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Ronellenfitsch, MD, Principal Investigator — Medical Faculty of the Martin Luther University Halle-Wittenberg
Locations (2):
- Germany (2):
  - University Hospital Carl Gustav Carus Dresden, Dresden, Saxony
  - University Hospital, Dpt. of Abdominal, Vascular and Endocrine Surgery, Halle

IPD SHARING:
Plan to Share IPD: Yes
In accordance with data protection regulations, individual de-identified individual participant data will be shared with other researchers upon reasonable and justified request. It is planned to store de-identified individual participant data on the B2SHARE repository of the EUDAT collaborative data infrastructure.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD will be made available after analysis of the primary outcome and after publication of pertaining results.
Access Criteria: Individual de-identified individual participant data will be shared with other researchers upon reasonable and justified request

REFERENCES:
- [Derived] Ronellenfitsch U, Kestel A, Klose J, Rebelo A, Bucher M, Ebert D, Mikolajczyk R, Wienke A, Kegel T, Hering J, Haiduk C, Richter M, Steighardt J, Grohmann E, Otto L, Kleeff J. Tranexamic Acid for reduction of intra- and postoperative TRansfusion requirements in elective Abdominal surgery (TATRA): study protocol for an investigator-initiated, multicenter, double-blind, placebo-controlled, randomized superiority trial with two parallel groups. Trials. 2024 Oct 19;25(1):695. doi: 10.1186/s13063-024-08541-8. PMID 39425234